CLINICAL TRIAL: NCT05758129
Title: Association Between PM2.5 Exposure and Nrf2-depended Ferroptosis Changes in Seizures Patients
Brief Title: Association Between PM2.5 Exposure and Ferroptosis in Seizures Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Affiliated Hospital of Jiangnan University (Other)
Responsible Party: Sponsor
Other Study IDs: 2022/11/16
Record Dates: First submitted 2023-02-11; First posted 2023-03-07 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-02

CONDITIONS: Exposure to Polluted Air
Keywords: PM2.5; seizures; IL-6; Nrf2; ferroptosis
MeSH Terms: conditions — Seizures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The control group: the invited recently diagnosed with epilepsy (< 2 months) live in Wuxi, Jiangsu, China (low PM2.5 level based on previous official PM2.5 records)
- The PM2.5 exposure group: the invited recently diagnosed with epilepsy live in Xuzhou, Jiangsu, China (high PM2.5 level based on previous official PM2.5 records)

SUMMARY:
This cohort study aims to discover the possible effects of PM2.5 exposures on the Nrf2- dependent ferroptosis pathway in seizure patients. This observational cohort's main question is whether PM2.5 exposures will affect the Nrf2- dependent ferroptosis pathway in seizure patients.

Participants will be divided into two groups: the control group and the air pollution to detect the biomarkers of the Nrf2- dependent ferroptosis pathway in seizure patients

DETAILED DESCRIPTION:
Background: Despite the exact mechanism of the effects of air pollution (PM2.5) on the central nervous system is still under debate. There is increasing evidence that air pollution (PM2.5) will affect neurodegenerative diseases including epilepsy. It is well known that air pollution (PM2.5) will increase the level of proinflammatory cytokine released by microglia, and advanced research indicated the level of interleukin-6 will affect epilepsy symptoms. In addition, our previous research indicated that Nrf2 plays a crucial role in seizure symptoms and cognitive function (NCT05269901). However, whether PM2.5-induced proinflammatory cytokine released by microglia will change Nrf2- dependent ferroptosis to facilitate seizure symptoms and cognitive function is still unexplored. Therefore, this pilot cohort study aims to discover the potential association between PM2.5 exposures and the changes in the interleukin-6 level and Nrf2- dependent ferroptosis pathway

Methods:

1. The investigators first enrolled 30 low PM2.5 exposure epileptic children and aged-matched high PM2.5 exposure children who were recently diagnosed with epilepsy (< 2 months)from two cities (Yangzhou and Xuzhou) as the control and air pollution group based on previous PM2.5 records;
2. Recorded the PM2.5 level in two cities every 5 days between 2022.12 and 2023.3 to compare the difference;
3. Interleukin-6 ELISA（IL6） KIT was used to compare the proinflammatory cytokine level in two groups
4. 4 Hydroxynonenal （4HNE） ELISA KIT was used to compare the lipid reactive oxygen species level in two groups
5. Real-Time Quantitative PCR（RT-qPCR） was used to compare messenger RNA (mRNA) expression of the Nrf2-dependent ferroptosis pathway (Nrf2, SLC7A11, GPX4) Detailed Methods protocol

1. PM2.5 level source: the PM2.5 levels were recorded via the data from the Ministry of Ecology and Environment of the People's Republic of China (air.cnemc.cn:18007/) 2. Sample collection: At the end of this study, the enrolled participant will come to the hospital to collect peripheral Blood (Affiliated Hospital of Jiangnan University and Xuzhou Children's Hospital, respectively), and the blood samples were collected into ethylene diamine tetraacetic acid（EDTA） vacutainer tubes and then divided into leukocytes and plasma for further experiments 3. Interleukin-6 and 4HNE: Plasma IL-6 and 4HNE concentrations were detected by the competitive ELISA method 4. RTqPCR sequence: h-GPX4 forward: 5'-GAGGCAAGACCGAAGTAAACTAC-3' h-GPX4 reverse: 5'-CCGAACTGGTTACACGGGAA-3' h-SLC7A11 forward: 5'-TCTCCAAAGGAGGTTACCTGC-3' h-SLC7A11 reverse: 5'-AGACTCCCCTCAGTAAAGTGAC-3' h-Nrf2 forward5'-ATAGCTGAGCCCAGTATC-3' h-Nrf2 reverse 5'- CATGCACGTGAGTGCTCT-3' h-GAPDH forward: 5'-GGAGCGAGATCCCTCCAAAAT-3' h-GAPDH reverse: 5'-GGCTGTTGTCATACTTCTCATGG-3'

ELIGIBILITY:
Inclusion Criteria:

1. Recently diagnosed with epilepsy (< 2 months)
2. living in this city for more than two years
3. no exposure to any chemistry pollution before

Exclusion Criteria:

1. abnormal IL-6 level before starting this pilot cohort
2. other neurological disorders except for epilepsy;
3. endocrine diseases;
4. cancer
5. receive anti-proinflammatory cytokines therapy

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The control group will be selected from the invited epileptic children who live in Wuxi city via the website, email, and poster. The PM2.5 group will be selected from the invited volunteers who live in Xuzhou city via the website, email, and poster.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-03-10 (Estimated); Study Completion 2023-03-25 (Estimated)

PRIMARY OUTCOMES:
The level changes of baseline IL6 three months later | From the date of all participants documented baseline data, until the date of the last participant documented the changes of biomarkers in peripheral blood, assessed up to 90 days
  Biomarkers of proinflammatory cytokine
The level changes of baseline 4HNE three months later | From the date of all participants documented baseline data, until the date of the last participant documented the changes of biomarkers in peripheral blood, assessed up to 90 days
  Biomarkers of ferroptosis, an indicator of lipid reactive oxygen species
The level changes of baseline of mRNA expression of the Nrf2-dependent ferroptosis three months later | From the date of all participants documented baseline data, until the date of the last participant documented the changes of biomarkers in peripheral blood, assessed up to 90 days
  Biomarkers of the Nrf2- dependent ferroptosis

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Hospital of JiangNan University, Department of Pediatrics, Wuxi, Jiangsu, China